CLINICAL TRIAL: NCT04141826
Title: Absorption of Peptides, Fluid, and Electrolytes in Patients With an Ileostomy
Acronym: ABSOLYT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Hvas (Other)
Responsible Party: Sponsor-Investigator, Christian Hvas, Consultant, associate professor, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-111-19
Record Dates: First submitted 2019-10-03; First posted 2019-10-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Nutritional Deficiency; Ileostomy; Functional Disturbance; Short Bowel Syndrome; Absorption; Disorder, Protein
MeSH Terms: conditions — Malnutrition; Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Production in separate facility, randomisation key kept by third party
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrolysed whey (Experimental): Hydrolysed whey
  Interventions: Dietary Supplement: Hydrolysed whey
- Intact whey (Active Comparator): Intact whey
  Interventions: Dietary Supplement: Intact whey
- Caseinate (Placebo Comparator): Caseinate
  Interventions: Dietary Supplement: Caseinate

INTERVENTIONS:
Dietary Supplement: Hydrolysed whey — 500 mL solution of 25 gram hydrolysed whey per day during 4 weeks
  Arms: Hydrolysed whey
Dietary Supplement: Intact whey — 500 mL solution of 25 gram intact whey per day during 4 weeks
  Arms: Intact whey
Dietary Supplement: Caseinate — 500 mL solution of 25 gram casein ate per day during 4 weeks
  Arms: Caseinate

SUMMARY:
Clinical trial, active comparator, cross over, randomised. In total, 12 adults with an ileostomy will be randomised to a sequential 4 weeks intervention with different qualities and sources of protein wish 2-week washout periods. Primary outcome: Ileostomy output.

DETAILED DESCRIPTION:
Patients with an ileostomy may be dehydrated and have nutritional deficiencies secondary to malabsorption of fluid, electrolytes, and nutrients. In this randomised, double blinded, crossover intervention study we aim to investigate how different protein sources affect intestinal absorption in patients with an ileostomy and intestinal insufficiency. Three oral solutions with different protein sources (hydrolysed whey, whey, and casein) will be administered in three different four-week intervention periods. The results will facilitate improved counselling and treatment of patients with an ileostomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old), male or female patients with an ileostomy and intestinal insufficiency
* Episodical or chronic sodium depletion defined by two urine samples with sodium levels ≤ 20 mmol/L, sampled with at least 28 days apart
* Six months or more after most recent bowel surgery
* If inflammatory bowel disease, no clinical signs of activity (any treatment allowed except systemic steroids > 10 mg/day)

Exclusion Criteria:

* Parenteral nutrition or intravenous fluid support ≥ 4000 mL/month
* Ongoing infection (C-reactive protein above 8 mg/L or core temperature >38.0°C)
* Self-reported intolerance to dairy products, including lactose intolerance
* Inability to understand Danish or the trial procedures
* Known or anticipated pregnancy
* Known severe renal insufficiency (eGFR < 20 mL/min)
* Known diabetes mellitus (HbA1c ≥ 48 mmol/mol (6.5%))
* Pacemaker, cochlear implants, or other electrical implants excludes the participants from BIA-measurements and measurements of GITT with 3D-Transit capsules, but not the remaining investigations
* Known intestinal stenosis or parastomal hernia excludes measurements of GITT with 3D-Transit capsules, but not the remaining investigations
* Abdominal diameter > 140 cm, or planned MR scan four weeks following participation excludes measurements of GITT with 3D-Transit capsules, but not the remaining investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
24-hour fecal wet weight | 4 weeks
  Difference in mean ileostomy output (wet weight) during 24 hours at the end of each intervention period

SECONDARY OUTCOMES:
Diuresis | 4 weeks
  24 hour urine volume
Natriuresis | 4 weeks
  24 hour urine sodium excretion
Amino acid absorption | 6 hours
  Plasma amino acids
Gastric and small bowel emptying | 6 hours
  3D transit evaluation
GLP1 and GLP2 | 6 hours
  Intestinal hormones during absorption
Portosystemic hepatic encephalopathy (PSE) test score, median value | 4 weeks
  Pen and paper test, score with range
Portosystemic hepatic encephalopathy (PSHE) test score abnormal (<4) | 4 weeks
  Pen and paper test, score with range
Continuous reaction time (CRT) index median | 4 weeks
  Reaction to 150 sound stimuli, read-out as index compared to normal values
Physical activity | 4 weeks
  Telemetric sensor
Body weight (kg) | 4 weeks
  Bio-impedance analysis (SECA)
Total body water (L) | 4 weeks
  Bio-impedance analysis (SECA)
Extracellular water (L) | 4 weeks
  Bio-impedance analysis (SECA)
Skeletal muscle mass (kg) | 4 weeks
  Bio-impedance analysis (SECA)
Fat-free mass (kg) | 4 weeks
  Bio-impedance analysis (SECA)
Fat mass (kg) | 4 weeks
  Bio-impedance analysis (SECA)

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Hvas, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data or selections herof will be shared upon specific agreements and with researchers who have legitimate causes, following contact to the PI
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: upon request, after publication
Access Criteria: contact to PI

REFERENCES:
- [Derived] Rud CL, Hvistendahl MK, Langdahl B, Kraglund F, Baunwall SMD, Lal S, Jeppesen PB, Hvas CL. Protein-based oral rehydration solutions for patients with an ileostomy: A randomised, double-blinded crossover study. Clin Nutr. 2024 Jul;43(7):1747-1758. doi: 10.1016/j.clnu.2024.05.038. Epub 2024 May 28. PMID 38850996